CLINICAL TRIAL: NCT05046834
Title: Investigation of the Effect of Cold Application on Patient's Pain and Vital Signs During Chest Tube Removal.
Brief Title: Effect of Cold Application on Patient's Pain and Vital Signs During Chest Tube Removal.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Researchers' workload and the fact that they work at different institutions made it difficult to gather data.
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Gonca Karayagiz Muslu, Associate professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 272
Record Dates: First submitted 2021-09-15; First posted 2021-09-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-07

CONDITIONS: Chest Tube Removal
Keywords: Chest Tube Removal, cold application, pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- cold application Group (Experimental): a cold gel pack will be wrapped in gauze and placed directly on the skin in an area with a radius of about 5 cm to cover the chest tube. The cold gel package will remain on the skin surface for about 20 minutes.
  Interventions: Other: cold application
- Cold Application Group with Thermometer (Experimental): 10 of cold application. After a minute, the skin temperature will be measured with an infrared thermometer if the temperature has dropped below 13.6 o C, the procedure will be terminated. If the skin temperature has not decreased below 13.6 0 C, the application will be continued, the application will be terminated when the temperature drops below the specified temperature.
  Interventions: Other: cold application until 13.6 C
- control Group (No Intervention): standard pain procedure.

INTERVENTIONS:
Other: cold application — Oral paracetamol 10 mg/kg, which is administered as standard 60 minutes before the procedure, will be given to patients who have decided to remove the chest tube by the physician and comply with the limitations of the study. After that, initial pain severity and vital signs of the patient will be recorded using FLACC 15 minutes before the start of the chest tube removal process (1.MEASURE). After this measurement, the cold gel package will be wrapped in gauze and placed directly on the skin, covering the area around the chest tube with a radius of about 5 cm. The cold gel package will remain on the skin surface for about 20 minutes. After 15 minutes, the cold package will be removed and the chest tube will be removed by the doctor.
  Arms: cold application Group
Other: cold application until 13.6 C — After measurements, the cold gel package, which rotates with one end open and forms a circle, will be wrapped in gauze and placed directly on the skin in a radius of about 5 cm, covering around the chest tube. 10 of the app. After the minute, the skin temperature will be measured with an infrared thermometer if the heat falls below 13.6 o C, the process will be terminated. If the skin temperature does not fall below 13.6 0 C, the application will continue, the application will be terminated when the heat falls below the specified temperature. After the cold package is removed, the chest tube will be removed by the doctor.
  Arms: Cold Application Group with Thermometer

SUMMARY:
In this study, the effect of cold application used during and after chest tube removal on pain and vital signs in infants and children in the 0-3 age group will be examined.

DETAILED DESCRIPTION:
Purpose of the research:In this study, the effect of cold application used during and after breast tube removal on pain and life signs in infants and children aged 0-3 years will be examined.

Hypotheses:

H1: children who have cold application around the tube 15 minutes before chest tube removal have low pain scores during chest tube removal compared to other groups.

H2: Children whose skin temperature is lowered below 13.60 C before breast tube removal have lower pain scores compared to other groups.

H3: The cold application technique in the group of children affects the crying time after the procedure.

H4: The cold application technique in the group of children affects the signs of life before and after the procedure.

The research is a study in randomized controlled, prospective and cross-sectional design.

The data of the study will be collected using the Patient Identification Information Form, FLACC Pain Scale, Life Signs Follow-up Form.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 0-3 years old,
* The chest tube is located for at least 24 hours,
* Without Mechanical ventilation support,
* Does not have any allergies to the drug
* Stable from the cardiovascular side

Exclusion Criteria:

* Children with any neurological diseases,
* Children with anynephrological
* Children with any respiratory diseases

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2026-10-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Pain assessed by FLACC | before cold application,
  the intensity of pain at the chest tube
Pain assessed by FLACC | immediately after chest tube removal ,
  the intensity of pain at the chest tube
Pain assessed by FLACC | 15 minutes after chest tube removal
  the intensity of pain at the chest tube
vital signs | before cold application,
  pulse, oxygen saturation, temperature, respiratory rate.
vital signs | immediately after chest tube removal ,
  pulse, oxygen saturation, temperature, respiratory rate.
vital signs | 15 minutes after chest tube removal
  pulse, oxygen saturation, temperature, respiratory rate.

SECONDARY OUTCOMES:
crying time | immediately after chest tube removal ,
  crying time because of pain (SECOND)
crying time | 15 minutes after chest tube removal
  crying time because of pain. (SECOND)

CONTACTS AND LOCATIONS:
Overall Officials: gonca muslu, Principal Investigator — Muğla Sıtkı Koçman University; dilek beytut, PhD, Study Chair — KKTC Lefke Europe University; saime yıldırım, nurse, Study Chair — Dr. Behçet Uz Child hospital; recep kara, PhD student, Study Chair — Muğla Sıtkı Koçman University; figen koyuncu, nurse, Study Chair — Dr. Behçet Uz Child hospital
Locations (1):
- Gonca Muslu, Fethiye, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No